CLINICAL TRIAL: NCT03230890
Title: HIRREM for Mitigation of PTSD Symptoms in Military Personnel
Brief Title: HIRREM in Military Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Brain State Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00028990
Record Dates: First submitted 2017-07-24; First posted 2017-07-27 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-10

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD; military; neurotechnology; HIRREM; allostasis; heart rate variability; baroreflex sensitivity; closed loop; acoustic stimulation; neural oscillations; autonomic; hyperarousal
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Single site, non-randomized, single arm, open label design,with collection of outcome measures before, and at intervals after the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- HIRREM (Experimental): This is the intervention, treatment arm that all participants receive in this open label, single arm trial. The intervention is High-resolution, relational, resonance-based, electroencephalic mirroring (HIRREM).
  Interventions: Device: HIRREM

INTERVENTIONS:
Device: HIRREM — HIRREM is a closed-loop, allostatic, acoustic stimulation neurotechnology intended to support auto-calibration of neural oscillations. The core technology is commercially available as a technique for relaxation. Scalp sensors monitor brain frequencies and amplitudes, and in real time, software algorithms translate specific frequencies into audible tones of varying pitch. These are reflected via earbuds in as little as 4-8 milliseconds. The in-office intervention for this study is administered as a series of up to twenty four, typically 1.5-2 hours sessions, comprised of 4-10 protocols (some eyes open, some eyes closed), lasting 6-40 minutes each, working at different scalp locations. Sessions are received over 12 days. Two sessions can be done in a half day. The intervention is received while comfortably seated in a zero gravity chair.

SUMMARY:
The purpose of this study is to evaluate the effects associated with the use of in-office High-resolution, relational, resonance-based, electroencephalic mirroring (HIRREM) for participants with symptoms of military-related traumatic stress. This is a single site, non-randomized, open label pilot study. Outcome measures collected before, and after the intervention evaluate effects on self-reported symptoms, autonomic cardiovascular regulation, functional measures, blood and saliva biomarkers of stress and inflammation, and network connectivity on whole brain, rest MRI testing. Self-reported symptom outcomes will also be collected remotely at 1, 3, and 6 months after completion of intervention. The study will assess feasibility in this cohort, focused on the Special Operations community, will provide estimates of effect size, and durability of symptom changes, while providing important pilot data for future proposals and investigations.

DETAILED DESCRIPTION:
This will be an open label, single site, pilot, clinical research study. Up to 40 active duty military personnel, or recent Veterans, age 18 or older, who have been diagnosed with PTSD, have received treatment for, are referred by military medical personnel for, or have active symptoms of military-related traumatic stress, with or without mild TBI, will be recruited to receive up to 24 HIRREM sessions over 2 weeks. For those who self-refer, and do not have a prior diagnosis or treatment for PTSD, active symptoms will be identified by a screening PCL-M score of 50 or greater. Recruitment of 40 participants will allow us to achieve the goal of 36 participants to complete the intervention, allowing for the possibility of dropouts. The primary outcome will be differential change in the PCL-M from baseline to completion of HIRREM sessions. Secondary measures include the Insomnia Severity Index (ISI), the Center for Epidemiological Studies Depression Scale (CES-D), an anxiety measure (GAD-7), a quality of life measure (EQ-5D), an autonomic symptom measure (Compass 31), and a daily sleep diary, as well as physiological measures including heart rate (HR), and blood pressure (BP), with calculation of heart rate variability measures (HRV), and baroreflex sensitivity (BRS). Functional measures will include reaction time (drop-stick paradigm), and grip strength (hydraulic dynamometer), and analysis of brain patterns. If there is a history of TBI, a Rivermead Post-Concussion Symptoms Questionnaire (RPQ) will be added. There will be pre- and post-intervention data collection for all measures (baseline, V1, and at completion of HIRREM sessions, V2). Self-report measures will also be repeated by phone at 1, 3, and 6 months after completion of sessions (V3, V4, and V5 respectively). The online sleep diary will be maintained from V1 until V3. A brainwave assessment will be obtained at V1.

ELIGIBILITY:
Inclusion Criteria:

Active duty military personnel, or recent veterans (Operation Enduring Freedom, Operation Iraqi Freedom, or Operation New Dawn), men and women, with a diagnosis of PTSD, or active symptoms suggesting PTSD as identified by a screening PCL-M score of 50 or greater, with or without traumatic brain injury (TBI), are eligible to participate in the study.

Exclusion Criteria:

* Unable, unwilling, or incompetent to provide informed consent
* Physically unable to come to the study visits, or to sit in a chair for several hours
* Known seizure disorder
* Severe hearing impairment (because the subject will be using ear buds during HIRREM)
* Ongoing need for treatment with opiate, benzodiazepine, or anti-psychotic medications, anti-depressant medications (SSRI, or SNRI's), sleep medications such as zolpidem or eszopiclone, stimulants such as Adderall, Provigil, or Ritalin, or thyroid hormone
* Anticipated and ongoing use of recreational drugs, alcohol, or energy drinks
* Lack of internet or smart phone access (will maintain remote access daily sleep diary through 1 month post-HIRREM visit)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-02-16 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles H Tegeler, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tegeler CH, Cook JF, Tegeler CL, Hirsch JR, Shaltout HA, Simpson SL, Fidali BC, Gerdes L, Lee SW. Clinical, hemispheric, and autonomic changes associated with use of closed-loop, allostatic neurotechnology by a case series of individuals with self-reported symptoms of post-traumatic stress. BMC Psychiatry. 2017 Apr 19;17(1):141. doi: 10.1186/s12888-017-1299-x. PMID 28420362
- [Background] Tegeler CH, Tegeler CL, Cook JF, Lee SW, Gerdes L, Shaltout HA, Miles CM, Simpson SL. A Preliminary Study of the Effectiveness of an Allostatic, Closed-Loop, Acoustic Stimulation Neurotechnology in the Treatment of Athletes with Persisting Post-concussion Symptoms. Sports Med Open. 2016 Dec;2(1):39. doi: 10.1186/s40798-016-0063-y. Epub 2016 Sep 14. PMID 27747793
- [Background] Fortunato JE, Tegeler CL, Gerdes L, Lee SW, Pajewski NM, Franco ME, Cook JF, Shaltout HA, Tegeler CH. Use of an allostatic neurotechnology by adolescents with postural orthostatic tachycardia syndrome (POTS) is associated with improvements in heart rate variability and changes in temporal lobe electrical activity. Exp Brain Res. 2016 Mar;234(3):791-8. doi: 10.1007/s00221-015-4499-y. Epub 2015 Dec 8. PMID 26645307
- [Background] Gerdes L, Tegeler CH, Lee SW. A groundwork for allostatic neuro-education. Front Psychol. 2015 Aug 17;6:1224. doi: 10.3389/fpsyg.2015.01224. eCollection 2015. PMID 26347688
- [Background] Tegeler CH, Shaltout HA, Tegeler CL, Gerdes L, Lee SW. Rightward dominance in temporal high-frequency electrical asymmetry corresponds to higher resting heart rate and lower baroreflex sensitivity in a heterogeneous population. Brain Behav. 2015 Jun;5(6):e00343. doi: 10.1002/brb3.343. Epub 2015 May 1. PMID 26085968
- [Background] Tegeler CH, Tegeler CL, Cook JF, Lee SW, Pajewski NM. Reduction in menopause-related symptoms associated with use of a noninvasive neurotechnology for autocalibration of neural oscillations. Menopause. 2015 Jun;22(6):650-5. doi: 10.1097/GME.0000000000000422. PMID 25668305
- [Background] Lee SW, Gerdes L, Tegeler CL, Shaltout HA, Tegeler CH. A bihemispheric autonomic model for traumatic stress effects on health and behavior. Front Psychol. 2014 Aug 1;5:843. doi: 10.3389/fpsyg.2014.00843. eCollection 2014. PMID 25136325
- [Background] Gerdes L, Gerdes P, Lee SW, H Tegeler C. HIRREM: a noninvasive, allostatic methodology for relaxation and auto-calibration of neural oscillations. Brain Behav. 2013 Mar;3(2):193-205. doi: 10.1002/brb3.116. Epub 2013 Jan 14. PMID 23532171
- [Derived] Tegeler CL, Gerdes L, Shaltout HA, Cook JF, Simpson SL, Lee SW, Tegeler CH. Successful use of closed-loop allostatic neurotechnology for post-traumatic stress symptoms in military personnel: self-reported and autonomic improvements. Mil Med Res. 2017 Dec 22;4(1):38. doi: 10.1186/s40779-017-0147-0. PMID 29502530

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HIRREM
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HIRREM
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.72 (6.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Change in PCL-M Score From Baseline to 12 Days
Description: The PTSD Checklist (PCL) - Military (M) is a symptom checklist to measure stress severity due to a traumatic experience in military settings. The PCL-M measures the American Psychiatric Association's Diagnostic and statistical manual of mental disorders (DSM-IV) of PTSD symptoms based on traumatic life experience. Seventeen items are rated on a Likert scale from 1 (not at all) to 5 (extremely), with a total score ranging from 17 to 85. Higher scores suggest more PTSD symptoms. Primary outcome for this pilot study will be change in PCL-M score from baseline to the immediate post-intervention in-person data collection at the completion of the HIRREM intervention (up to 12 days later).
Time Frame: Data is collected at baseline and immediately following completion of the HIRREM intervention (up to 12 days later)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIRREM
Number analyzed (Participants) | 32
score on a scale | -12.88 (9.11)

2. Secondary Outcome: Change in Center for Epidemiologic Studies Depression Scale (CES-D) Score From Baseline to 12 Days
Description: The CES-D is a 20-item survey assessing affective depressive symptomatology to screen for risk of depression. Scores range from 0-60, with a score of 16 commonly used as a clinically relevant cut-off. Higher scores suggest more depressive symptomatology. Secondary outcome with the CES-D will be analyzed for change from baseline to the immediate post-HIRREM in person data collection.
Time Frame: Data is collected at baseline and immediately following completion of the intervention (up to 12 days later)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HIRREM
Number analyzed (Participants) | 32
units on a scale | -13.69 (9.24)

3. Secondary Outcome: Change in Insomnia Severity Index (ISI) Score From Baseline to 12 Days
Description: The severity of insomnia symptoms is measured using the ISI with each data collection visit. The ISI is a 7 question measure, with responses from 0-4 for each question, yielding scores ranging from 0-28. Higher scores indicate the strength of the insomnia severity. Secondary outcome with the ISI will be analyzed for change from baseline to the immediate post-HIRREM in person data collection.
Time Frame: Data is collected at baseline and immediately following completion of the intervention (up to 12 days later)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIRREM
Number analyzed (Participants) | 32
score on a scale | -6.31 (5.03)

4. Secondary Outcome: Change in Generalized Anxiety Disorder-7 (GAD-7) Score From Baseline to 12 Days
Description: The Generalized Anxiety Disorder-7 (GAD-7) is a seven item screening tool for anxiety that is widely used in primary care. Each item is rated from 0 (not at all) to 3 (nearly every day). Scores range from 0 to 21 with higher scores suggesting more anxiety. Secondary outcome with the GAD-7 will be analyzed for change from baseline to the immediate post-HIRREM in person data collection.
Time Frame: Data is collected at baseline and immediately following completion of the intervention (up to 12 days later)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIRREM
Number analyzed (Participants) | 32
score on a scale | -6.69 (4.72)

5. Secondary Outcome: Change in Rivermead Post-Concussion Symptoms Questionnaire (RPQ) Score From Baseline to 12 Days
Description: The Rivermead Post-Concussion Symptoms Questionnaire (RPQ) is a 16-item survey that assesses the severity of the most common post-concussion symptoms on a scale of 0 to 4, with a total score range from 0 to 64 (least to greatest symptom severity). Items are compared to levels before the head injury and are reported as a 24 hour recall. Secondary outcome with the RPQ will be analyzed for change from baseline to the immediate post-HIRREM in person data collection.
Time Frame: Data is collected at baseline and immediately following completion of the intervention (up to 12 days later)
Population: Two participants did not have history of concussion and did not complete measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIRREM
Number analyzed (Participants) | 30
score on a scale | -10.70 (11.71)

6. Secondary Outcome: Change in EQ-5D Score From Baseline to 12 Days
Description: The EQ-5D is a brief, standardized measure of health status developed by the EuroQol Group, and is a paper and pencil survey providing a single index value for health status. Secondary outcome with the EQ-5D will be analyzed for change from baseline to the immediate post-HIRREM in person data collection. Global health rating question is reported (0-100, with 100 being in the best health possible).
Time Frame: Data is collected at baseline and immediately following completion of the intervention (up to 12 days later)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIRREM
Number analyzed (Participants) | 32
score on a scale | 9.59 (12.35)

7. Secondary Outcome: Change in Heart Rate Variability Measure of SDNN From Baseline to 12 Days
Description: Secondary autonomic outcome with heart rate variability will be analyzed for change from baseline to the immediate post-HIRREM in person data collection. Heart rate variability is measured in the time domain as standard deviation beat-to-beat interval (SDNN, milliseconds). For calculation of SDNN, the R-R intervals are visually inspected, and data considered as artifact is manually removed. Higher SDNN values suggest better autonomic regulation.
Time Frame: Data is collected at baseline and immediately following completion of the intervention (up to 12 days later)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | HIRREM
Number analyzed (Participants) | 32
ms | 9.43 (17.43)

8. Secondary Outcome: Change in Baroreflex Sensitivity HF Alpha From Baseline to 12 Days
Description: Blood pressure and heart rate are acquired from 10 minute recordings of noninvasive finger arterial pressure measurements and ECG with participants lying quietly, supine. Systolic BP and beat to beat, RR intervals files generated via the data acquisition system (BIOPAC acquisition system and Acknowledge 4.2 software, Santa Barbara, CA), at 1000 Hz, are analyzed using Nevrokard Baroreflex Sensitivity (BRS) software (Nevrokard BRS, Medistar, Ljubljana, Slovenia). Analysis is conducted on the first complete 5-minute epoch that is considered to be acceptable for analysis. Evaluation includes analysis for measures of spontaneous baroreflex sensitivity (BRS), in the frequency domain as high frequency (HF) alpha index (ms2). Secondary autonomic outcome with BRS will be analyzed for change from baseline to the immediate post-HIRREM in person data collection. Higher values in HF alpha suggest better autonomic regulation.
Time Frame: Data is collected at baseline and immediately following completion of the intervention (up to 12 days later)
Measure: Mean (Standard Deviation); unit: ms2
Arm/Group | HIRREM
Number analyzed (Participants) | 32
ms2 | 9.43 (12.05)

9. Secondary Outcome: Change in Baroreflex Sensitivity Sequence Up From Baseline to 12 Days
Description: Blood pressure and heart rate are acquired from 10 minute recordings of noninvasive finger arterial pressure measurements and ECG with participants lying quietly, supine. Systolic BP and beat to beat, RR intervals files generated via the data acquisition system (BIOPAC acquisition system and Acknowledge 4.2 software, Santa Barbara, CA), at 1000 Hz, are analyzed using Nevrokard Baroreflex Sensitivity (BRS) software (Nevrokard BRS, Medistar, Ljubljana, Slovenia). Analysis is conducted on the first complete 5-minute epoch that is considered to be acceptable for analysis. Evaluation includes analysis for measures of spontaneous baroreflex sensitivity (BRS), in the time domain as frequency domain as BRS Sequence Up (ms/mmHg). Secondary autonomic outcome with BRS will be analyzed for change from baseline to the immediate post-HIRREM in person data collection. Higher values in Sequence Up suggest better autonomic regulation.
Time Frame: Data is collected at baseline and immediately following completion of the intervention (up to 12 days later)
Measure: Mean (Standard Deviation); unit: ms/mmHg
Arm/Group | HIRREM
Number analyzed (Participants) | 32
ms/mmHg | 7.46 (12.33)

10. Secondary Outcome: Change in Baroreflex Sensitivity Sequence Down From Baseline to 12 Days
Description: Blood pressure and heart rate are acquired from 10 minute recordings of noninvasive finger arterial pressure measurements and ECG with participants lying quietly, supine. Systolic BP and beat to beat, RR intervals files generated via the data acquisition system (BIOPAC acquisition system and Acknowledge 4.2 software, Santa Barbara, CA), at 1000 Hz, are analyzed using Nevrokard Baroreflex Sensitivity (BRS) software (Nevrokard BRS, Medistar, Ljubljana, Slovenia). Analysis is conducted on the first complete 5-minute epoch that is considered to be acceptable for analysis. Evaluation includes analysis for measures of spontaneous baroreflex sensitivity (BRS), in the time domain as frequency domain as BRS Sequence Down (ms/mmHg). Secondary autonomic outcome with BRS will be analyzed for change from baseline to the immediate post-HIRREM in person data collection. Higher values in Sequence Down suggest better autonomic regulation.
Time Frame: Data is collected at baseline and immediately following completion of the intervention (up to 12 days later)
Measure: Mean (Standard Deviation); unit: ms/mmHg
Arm/Group | HIRREM
Number analyzed (Participants) | 32
ms/mmHg | 5.56 (9.16)

11. Secondary Outcome: Change in Baroreflex Sensitivity Sequence All From Baseline to 12 Days
Description: Blood pressure and heart rate are acquired from 10 minute recordings of noninvasive finger arterial pressure measurements and ECG with participants lying quietly, supine. Systolic BP and beat to beat, RR intervals files generated via the data acquisition system (BIOPAC acquisition system and Acknowledge 4.2 software, Santa Barbara, CA), at 1000 Hz, are analyzed using Nevrokard Baroreflex Sensitivity (BRS) software (Nevrokard BRS, Medistar, Ljubljana, Slovenia). Analysis is conducted on the first complete 5-minute epoch that is considered to be acceptable for analysis. Evaluation includes analysis for measures of spontaneous baroreflex sensitivity (BRS), in the time domain as frequency domain as BRS Sequence All (ms/mmHg). Secondary autonomic outcome with BRS will be analyzed for change from baseline to the immediate post-HIRREM in person data collection. Higher values in Sequence All suggest better autonomic regulation.
Time Frame: Data is collected at baseline and immediately following completion of the intervention (up to 12 days later)
Measure: Mean (Standard Deviation); unit: ms/mmHg
Arm/Group | HIRREM
Number analyzed (Participants) | 32
ms/mmHg | 5.75 (8.21)

12. Secondary Outcome: Change in Drop Stick Reaction Time From Baseline to 12 Days
Description: Reaction testing is measured by a drop-stick apparatus that has been validated as a way to quantify the impact of athletic concussion on psychomotor performance. Following two practice trials, participants perform eight trials, and a mean distance value is calculated. Secondary functional outcome with drop-stick reaction time will be analyzed for changes in distance from baseline to the in person data collection immediately after completion of the intervention. A lower average indicates a faster reaction time.
Time Frame: Data is collected at baseline and immediately following completion of the intervention (up to 12 days later)
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | HIRREM
Number analyzed (Participants) | 32
cm | -3.86 (6.64)

13. Secondary Outcome: Change in Grip Strength From Baseline to 12 Days
Description: Grip strength will evaluated using a hydraulic hand dynamometer (Baseline Hydraulic Hand Dynamometer, ranges from 0 to 300 lbs). Both right and left hand will be evaluated, and the greatest force generated during three trials will be used for analysis. A higher score indicates stronger grip strength.
Time Frame: Data is collected at baseline and immediately following completion of the intervention (up to 12 days later)
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | HIRREM
Number analyzed (Participants) | 32
lbs
  Right Hand | 1.74 (13.25)
  Left Hand | 1.94 (11.19)

14. Secondary Outcome: Change in Functional MRI From Baseline to 12 Days
Description: Anatomical and physiological brain imaging will be performed during a 1-hour imaging session at baseline and immediately following completion of the intervention. This will include imaging sequences such as high resolution structural scans. Brain network data will be collected using blood oxygenation level dependent (BOLD) scans. These scans will be collected under various states such as at rest. All images will be acquired using a 3 Tesla Siemens MRI scanner. Whole-brain network connectivity will be assessed using blood oxygenation level dependent (BOLD) imaging. Unit of measure is percentage of BOLD signal change. Community structure will be determined for each participant pre- and post-intervention. This project will focus on the community including the Default Mode Network (DMN). Participant strength of the community structure will be determined of the DMN. Permutation analysis will be used to evaluate significant pattern change in specific networks.
Time Frame: Data is collected at baseline and immediately following completion of the intervention (up to 12 days later)
Population: Due to funding limitations, only 18 received fMRI scans.
Measure: Mean (Standard Deviation); unit: % blood oxygenation level dep (BOLD)
Arm/Group | HIRREM
Number analyzed (Participants) | 18
% blood oxygenation level dep (BOLD) | -0.012 (0.034)

15. Secondary Outcome: Change in Blood Biomarkers for Stress and Inflammation Score From Baseline to 12 Days
Description: Blood for a panel of biomarkers for stress will be collected at enrollment, and after completion of the intervention. The panel includes Ang II, Ang 1-7, Epinephrine, Norepinephrine, C-reactive protein, Vasopressin, IL-1, IL-6, and IL-10.
Time Frame: Data is collected at baseline and immediately following completion of the intervention (up to 12 days later)
Population: Due to funding limitations, only 15 people received biomarker measures. One sample was unable to be used, so n=14 is presented.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | HIRREM
Number analyzed (Participants) | 14
pg/ml
  Ang II (pg/ml) | -0.50 (23.17)
  Ang 1-7 (pg/ml) | 5.11 (16.94)
  Epinephrine (pg/ml) | -5.87 (20.66)
  Norepinephrine (pg/ml) | -29.98 (165.88)
  Vasopressin (pg/ml) | -0.19 (0.77)
  IL-1 (pg/ml) | -0.20 (0.07)
  IL-6 (pg/ml) | -0.06 (0.21)
  IL-10 (pg/ml) | -0.09 (0.22)

16. Secondary Outcome: Salivary Biomarker Cortisol for Stress From Baseline to 12 Days
Description: Saliva for salivary biomarker Cortisol, for stress, will be collected at enrollment, and after completion of the intervention.
Time Frame: Salivary biomarker for stress will be obtained at baseline and immediately following completion of the intervention (up to 12 days)
Population: One participant had a bad file for salivary amylase (n=14).
Measure: Mean (Standard Deviation); unit: ug/dl
Arm/Group | HIRREM
Number analyzed (Participants) | 14
ug/dl | 0.04 (0.13)

17. Secondary Outcome: Change in Epigenetic Markers From Baseline to 12 Days
Description: DNA will be isolated from whole blood, collected in yellow-top Vacutainer tubes (ACD as the preservative), using the AutoPure LS system in the Genomics Center Core lab. DNA will be bisulfite-converted using the EZ DNA Methylation Gold kit (Zymo, Irvine, CA). To quantify DNA methylation at each site, investigators will use the HumanMethylationEPIC450 BeadChip (Illumina, Inc.). The methylation proportion for each site (beta value) is based on the ratio of the fluorescence intensity of the methylated versus the combined methylated & unmethylated probes, & will be determined with GenomeStudio (Illumina, Inc.). Ratio of 0 equals no methylation & ratio of 1 equals total (100%) methylation." Effects of DNA methylation for a specific site are dependent on function of the regulated gene(s). For some genes, increased level methylation from the intervention may be beneficial, while for others an increased level may be detrimental. There is no universal way to interpret change in DNA methylation.
Time Frame: Blood for epigenetic markers will be obtained at baseline and immediately following completion of the intervention (up to 12 days)
Population: Only a subset of the main cohort had this testing done due to limited funds.
Measure: Mean (Standard Deviation); unit: ratio of methylation
Arm/Group | HIRREM
Number analyzed (Participants) | 8
ratio of methylation | -.00038 (0.006003)

18. Secondary Outcome: Change in Sleep Latency Score From Baseline to 42 Days
Description: An online daily sleep diary to calculate sleep latency will be maintained from baseline, through the one month post-intervention remote data collection (roughly 42 days). Sleep latency is reported in minutes and a smaller score suggests falling asleep faster.
Time Frame: Sleep diary data will be collected daily via online access from baseline to a month following completion of intervention (up to 42 days)
Population: Due to initial funding, only the first 18 participants received the sleep diary.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | HIRREM
Number analyzed (Participants) | 18
minutes | 36.01 (27.24)

19. Secondary Outcome: Change in C-reactive Protein for Stress and Inflammation Score From Baseline to 12 Days
Description: Blood for biomarker C-reactive protein for stress will be collected at enrollment, and after completion of the intervention.
Time Frame: Data is collected at baseline and immediately following completion of the intervention (up to 12 days later)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | HIRREM
Number analyzed (Participants) | 14
mg/dl | -0.10 (0.19)

20. Secondary Outcome: Salivary Biomarker for Stress From Baseline to 12 Days
Description: Saliva for salivary biomarker Alpha-Amylase, for stress, will be collected at enrollment, and after completion of the intervention.
Time Frame: Salivary biomarker Alpha-Amylase for stress will be obtained at baseline and immediately following completion of the intervention (up to 12 days)
Population: One participant had a bad file for salivary amylase (n=14).
Measure: Mean (Standard Deviation); unit: (U/ml)
Arm/Group | HIRREM
Number analyzed (Participants) | 14
(U/ml) | 15.00 (16.66)

ADVERSE EVENTS:
Time Frame: Enrollment, immediately following completion of the intervention, and at later remote data collections 1, 3, and 6 months post-intervention.
Arm/Group | HIRREM
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT03230890/Prot_SAP_002.pdf
  • Informed Consent Form (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT03230890/ICF_003.pdf